CLINICAL TRIAL: NCT06940934
Title: ANCRAGE: Post-Market Product Surveillance of Intracranial ANeurysms Treated With Commercial ReGistered ACANDIS Devices in FrancE
Brief Title: Post-Market Product Surveillance of Intracranial ANeurysms Treated With Commercial ReGistered ACANDIS Devices in FrancE
Acronym: ANCRAGE PMS
Status: Recruiting | Type: Observational
Sponsor: Acandis GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: ANCRAGE PMS
Record Dates: First submitted 2025-04-16; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Intracranial Aneurysms
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Devices of the DERIVO family
- ACCLINO flex plus Stent

SUMMARY:
The aims of this clinical data collection are to investigate mortality, morbidity and neurological outcome 12 months after treatment of subject's intracranial aneurysm(s) and additionally to evaluate potential residual risks associated with the use of the commercial device(s) and to ensure the long-term safety and performance of Acandis Device(s) after its placing on the French market. On top of this, these cohorts will generate data for getting the renewal of the device's reimbursement on the French market.

ELIGIBILITY:
Inclusion Criteria:

* The subject has an intracranial aneurysm that can be treated with one of the Acandis device indicated for the treatment of intracranial aneurysms.
* The subject is 18 years of age or older.
* The subject is willing to comply with scheduled visits and examinations, per institution standard of care.

Exclusion Criteria:

* The subject has provided tacit opposition to data collection.
* Any IFU warning will be considered for exclusion in the cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Each cohort will consist of subjects with an intracranial aneurysm whom the physician wishes to treat with one or more Acandis devices.
  Each subject will be followed according to the standard of care within the participating sites.
  All treated (and intended to treat with at least 1 Acandis device inserted) cases will be captured in the ANCRAGE study database, from the date of agreement with French authorities; that means it will be a consecutive prospective enrollment to demonstrate the exhaustivity at the site, even the cases are captured in the database retrospectively.
  There is a minimum of 50 consecutive cases to be enrolled per device family, from the time the device has been put on the French market and until the needed report to the authorities (for instance the renewal of the device registration/reimbursement).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Morbi-mortality related to the device and/or procedure at 12+/-3 months post implantation | 12+/-3 months after treatment
  Morbi-mortality related to the device and/or procedure at 12+/-3 months post implantation, defined as a mRS >/= 3 for the subjects with a baseline mRS between 0 and 2 or mRS increase of 1 point for subjects with a baseline mRS greater than 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Neuroradiologie Interventionnelle, CHU de Rouen (Charles Nicolle), Rouen, France